CLINICAL TRIAL: NCT05188378
Title: A Phase 1, Randomized, Double-blind, Two-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics and Safety of Two Subcutaneous Injection Formulations of Tocilizumab (CT-P47 and EU-approved RoActemra) in Healthy Subjects
Brief Title: A Study to Compare the Pharmacokinetics and Safety of CT-P47 and RoActemra in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CT-P47 1.1
Record Dates: First submitted 2021-12-10; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-P47 (Experimental): 162 mg in 0.9 mL, a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: CT-P47
- EU-approved RoActemra (Active Comparator): 162 mg in 0.9 mL, a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Interventions: Biological: EU-approved RoActemra,

INTERVENTIONS:
Biological: CT-P47 — 162 mg in 0.9 mL, a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Arms: CT-P47
Biological: EU-approved RoActemra, — 162 mg in 0.9 mL, a single subcutaneous (SC) injection via pre-filled syringe (PFS)
  Arms: EU-approved RoActemra

SUMMARY:
A study to Compare the Pharmacokinetics and Safety of CT-P47 and RoActemra in Healthy Subjects

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio to receive a single dose (162 mg) of either CT-P47 or EU-approved RoActemra.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Body weight of ≥60 and ≤100 kg for male and ≥50 and ≤100 kg for female and a BMI between 18.5 and 28.0 kg/m2 (both inclusive) when rounded to the nearest tenth

Exclusion Criteria:

* A medical history and/or condition that is considered significant
* Clinically significant allergic reactions, hypersensitivity
* History or current infection of hepatitis B virus, hepatitis C virus, human immunodeficiency virus, or syphilis
* Active or latent Tuberculosis
* History of malignancy
* Previous exposure to tocilizumab or any drug that targets IL-6

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary objective | up to Day 43
  To demonstrate PK similarity in terms of Area under the zero to infinity (AUC0-inf)
Primary objective | up to Day 43
  To demonstrate PK similarity in terms of Area under the concentration-time curve from time zero to the last quantifiable concentration (AUC0-last)
Primary objective | up to Day 43
  To demonstrate PK similarity in terms of Maximum serum concentration (Cmax)

CONTACTS AND LOCATIONS:
Overall Officials: KyungSang Yu, Principal Investigator — Seoul National University Hospital; JaeYong Chung, Principal Investigator — Seoul National University Bundang Hospital; HyeWon Chung, Principal Investigator — Korea University Guro Hospital; DongSeong Shin, Principal Investigator — Gachon University Gil Medical Center; MinKyu Park, Principal Investigator — Chungbuk National University Hospital; MinGul Kim, Principal Investigator — Jeonbuk National University Hospital; JongLyul Ghim, Principal Investigator — Inje University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu KS, Kim B, Shin D, Park MK, Hwang JG, Kim MG, Chung H, Ghim J, Chung JY, Smolen JS, Burmester GR, Kim S, Bae Y, Jeon D, Yoo J, Yang G, Bae J, Keystone E. Pharmacokinetics and safety of candidate tocilizumab biosimilar CT-P47 versus reference tocilizumab: a randomized, double-blind, single-dose phase I study. Expert Opin Investig Drugs. 2023 May;32(5):429-439. doi: 10.1080/13543784.2023.2212155. Epub 2023 May 26. PMID 37231670